CLINICAL TRIAL: NCT03961048
Title: Ideal Initial Bolus and Infusion Rate for Erector Spinae Plane Block Catheters
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Change in hospital protocol
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HM20014242
Record Dates: First submitted 2019-05-21; First posted 2019-05-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Pain, Postoperative; Pain, Chest
Keywords: Erector Spinae; Cardiac Surgery; Regional Anesthesia
MeSH Terms: conditions — Pain, Postoperative; Chest Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Bilateral catheters (Experimental): patients receiving bilateral catheters (such as for patients undergoing sternotomies/midline incisions or with planned bilateral thoracotomy incisions)
  Interventions: Drug: Ropivacaine 0.2%-Sodium Chloride 0.9% Injectable Solution bilaterally
- Single catheter (Experimental): patients who only have one catheter in place (such as in patients who have unilateral thoracotomies and not midline sternotomies)
  Interventions: Drug: Ropivacaine 0.2%-Sodium Chloride 0.9% Injectable Solution unilaterally

INTERVENTIONS:
Drug: Ropivacaine 0.2%-Sodium Chloride 0.9% Injectable Solution bilaterally — Variable initial post-operative dose of 10cc to 40cc bilaterally with a variable programmed dose to be repeated afterward of 10cc to 40cc of 0.2% ropivacaine every 6 hours bilaterally.
  Arms: Bilateral catheters
Drug: Ropivacaine 0.2%-Sodium Chloride 0.9% Injectable Solution unilaterally — Variable initial post-operative dose of 10cc to 40cc unilaterally with a variable programmed dose to be repeated afterward of 10cc to 40cc of 0.2% ropivacaine every 6 hours unilaterally.
  Arms: Single catheter

SUMMARY:
This study would like to identify the best starting dose and infusion rate for nerve blocks and nerve catheters related to the erector spinae plane block that can improve functional status and pain control on cardiac surgery patients and minimize the necessity for opioid pain control using a continuous reassessment model.

DETAILED DESCRIPTION:
The study will continue taking steps in helping to identify the role erector spinae plane nerve blocks have in thoracic surgery. This is a relatively new nerve block (first identified and described in 2016) and the studies that have been done and the case series that have been reported have been very promising in supporting its role in thoracic surgery. As it is a plane block (not around a specific nerve but in a general area), larger volumes and doses often have to be used in these sorts of blocks (such as a transverses abdominalis plane block) to get good spread of the local anesthetic in the plane to reach the desired nerves that pass through this plane with one injection. Our hospital has been doing these blocks for patients as a standard of care for them, but this study will take a closer look to see if there is an optimal dose and volume of medicine to improve patients' functional status and pain control to minimize the need for opioids. The study will use a continuous reassessment model to determine the optimal dose.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing planned thoracotomies and sternotomies for cardiothoracic surgery who will be taken to the cardiac surgery ICU postoperatively

Exclusion Criteria:

* BMI >40
* infection at the proposed catheter site
* ongoing sepsis/bacteremia
* patient unable to sit up for the procedure
* patients requiring significant vasopressor support (>1 vasopressor)
* patient refusal
* less than 18 years of age (they are managed in the pediatric ICU rather than the Cardiac Surgery ICU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Median Effective Dose | 6.5 hours
  Dose at which 50% of patients achieve a clinically significant nerve block after a single bolus and after periodic programmed boluses of Ropivacaine as represented by either an adequate decrease in sensation of the chest (covering at least 5 dermatomes) or an improvement in vital capacity breaths (of 500 mL or more)

SECONDARY OUTCOMES:
Change in pain rating | From just before to 30 minutes after a bolus is administered
  Self reported pain rating on a 0-10 scale where 0 is no pain and 10 is pain as bad as it can be
Change in heart rate | From just before to 30 minutes after a bolus is administered
  Heart rate measured using a heart rate monitor
Blood pressure | From just before to 30 minutes after a bolus is administered
  Blood pressure measured using a blood pressure monitor
Change in percent oxygen saturation of hemoglobin | From just before to 30 minutes after a bolus is administered
  Pulse oximetry reading from a monitor
Changes in electrocardiogram tracing | From just before a bolus is administered to 6.5 hours
  Monitoring for changes in electrical conduction in the heart as monitored by the continuous 5 lead electrocardiogram tracing, watching for any side effects.
Dermatomal coverage | From just before to 30 minutes after a bolus is administered
  The area of numbness experienced in the chest wall as measured using a pinprick test and documented on a cartoon map showing a chest wall and dermatomal borders
Opioid consumption | 6.5 hours
  Total opioid medication consumption during the study period
Non-narcotic pain medication consumption | 6.5 hours
  Total non-narcotic pain medicine consumption during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Bryant Tran, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No